CLINICAL TRIAL: NCT00553904
Title: Long-Term Effects of Cranberry Juice on Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Effect of Cranberry Juice on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Joseph A. Vita, MD, Boston University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-26708
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Cranberry juice — 480 ml of double strength cranberry juice daily for four weeks

SUMMARY:
A pilot study of 15 subjects will be completed to determine whether acute consumption of cranberry juice has an effect on endothelial function. We will then complete a randomized, double blind, placebo controlled crossover study designed to investigate the effects of cranberry juice consumption on endothelial function. Participants (n=40) will drink 480 ml of double strength cranberry juice or a similar appearing and tasting placebo per day for four weeks. After a two week rest period, they will cross over to the other beverage. We will examine endothelial function before and after each of the two treatment periods. The study will provide information about the chronic vascular effects of cranberry juice.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease

Exclusion Criteria:

* Pregnant and lactating women
* Clinical history of other major illness including end-stage cancer, renal failure, hepatic failure, gastrointestinal disorders that may impair absorption, or other conditions that in the opinion of the principal investigator make a clinical study inappropriate
* Treatment with an investigational new drug within the last 30 days
* History of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Treatment with Vitamin E, Vitamin C, beta carotene, lipoic acid, or other food or herbal supplements within 2 weeks of enrollment (subjects taking multivitamins or other forms of vitamin E and C in doses that do not exceed two times the RDA will not be excluded).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 1 month

SECONDARY OUTCOMES:
Carotid-femoral pulse wave velocity | 1 month
Markers of inflammation | 1 month
Serum anthocyanins | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dohadwala MM, Holbrook M, Hamburg NM, Shenouda SM, Chung WB, Titas M, Kluge MA, Wang N, Palmisano J, Milbury PE, Blumberg JB, Vita JA. Effects of cranberry juice consumption on vascular function in patients with coronary artery disease. Am J Clin Nutr. 2011 May;93(5):934-40. doi: 10.3945/ajcn.110.004242. Epub 2011 Mar 16. PMID 21411615